CLINICAL TRIAL: NCT02725892
Title: LuCaReAl: Lung Cancer Registry in Algeria.
Brief Title: National Lung Cancer Registry in Men and Women Based on Diagnosis in Algeria
Acronym: LuCaReAl
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133FR00108
Record Dates: First submitted 2016-03-11; First posted 2016-04-01 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Oncology & Epidemiology & Lung Cancer
Keywords: lung cancer epidemiology algeria registry
MeSH Terms: conditions — Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 72 Months

GROUPS / COHORTS (1):
- lungcancer patients: Men or women diagnosed with lung cancer all types and stages confirmed over 12 months of recruitment period by a pathologist
  Interventions: Other: NIS observational stud

INTERVENTIONS:
Other: NIS observational stud — NIS observational study : Epidemiologic registry

SUMMARY:
National, prospective, multicentric, non-interventional registry-based study, conducted among oncologists, pulmonologists in community and university hospitals, from the public sector in Algeria.

The study will collect information on the characteristics, and lung carcinomas patterns of patients whose lung cancer diagnosis was confirmed by a pathologist during the study period.

DETAILED DESCRIPTION:
The study consists of:

* All patients meeting inclusion/exclusion criteria presenting to their oncologists/pulmonologists for a routine visit during recruitment period will be sequentially asked to participate to the study.
* The patients who do not consent will only be reported as new case of lung cancer for the incidence study.

The patients who consent to participate to the study will perform four in-hospital visits (Inclusion visit, visit at 3, 6 and 12 months). In addition to the 4 visits, a phone contact with the patients every 6 months at years 2,3, 4 and 5 will be done by the investigator or one of his/her authorised representative or the CRO or during a routine visit to the investigator, to check the patient's survival status.

THE STUDY DURATION 72 MONTHS

ELIGIBILITY:
Inclusion Criteria:

* Men or women diagnosed with lung cancer all types and stages confirmed over 12 months of recruitment period by a pathologist

  * Aged at least18 years at diagnosis
  * Patients who provide their informed consent form

Exclusion Criteria:

* Patients who did not provide the informed consent form
* Patients with a mental or psychological disorder according to their treating clinicians

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: each sanitary region defined by the Ministry of health, the investigational centres will propose to all patients whom met illegibility criteria to participate to the study.
  Whenever possible, comprehensive lists of hospitals will be used as a data source in the site selection process. Lists will be obtained either from national authorities, local scientific societies or professional associations, depending on the local availability of this type of information. All efforts will be made to approach and select sites/physicians for the present study if they can provide a representative sample.
  The formal sample size will be calculated among the representatives hospitals sites overall the country.
Sampling Method: Non-Probability Sample
Enrollment: 897 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
incidence of lung cancer | 12 months of recruitment period
  incidence of lung cancer, all types, stages and ages combined, in men and women newly diagnosed with lung cancer in Algeria over 12 months of recruitment period

SECONDARY OUTCOMES:
incidence of newly diagnosed lung cancer | 12 month period
  1) To characterise the incidence of newly diagnosed lung cancer in Algeria in a 12 month period according to patient and disease characteristics (Wilaya, sex, age, lung cancer type, stage disease and smoking status).
survival | at 12, 24, 36, 48 and 60 months of follow-up.
quality of life -EORTC QLQ-C30 | baseline, 3, 6 and 12 months follow-up.
  To evaluate the quality of life of patients diagnosed with lung cancer in Algeria according to EORTC QLQ-C30 )
Quality Of Life-EORTC QLQ- LC13 | baseline, 3, 6 and 12 months follow-up.
  To evaluate the quality of life of patients diagnosed with lung cancer in Algeria according to EORTC QLQ- LC13

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Bouzid, Principal Investigator — CPMC; Habib Douagui, respiratory Diseases, Principal Investigator — Beni messous
Locations (3):
- Algeria (3):
  - Research Site, Algiers
  - Research Site, Constantine
  - Research Site, Oran

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133FR00108&attachmentIdentifier=a710a0bc-7aec-4b11-9b83-219006bd9317&fileName=D133FR00108_Synopsis_Redacted.pdf&versionIdentifier=